CLINICAL TRIAL: NCT03142243
Title: Morphological Asymmetry in Elite Female Tennis Players Competing in an International Tournament in Belgium: an Observational Study
Brief Title: Morphological Asymmetry in Elite Female Tennis Players
Acronym: AsymFemaleTP
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Vrije Universiteit Brussel (Other)
Responsible Party: Principal Investigator, Laurent Chapelle, Researcher, Vrije Universiteit Brussel
Other Study IDs: Asym Female Elite TP
Record Dates: First submitted 2017-05-03; First posted 2017-05-05 (Actual); Last update posted 2017-05-19 (Actual); Status verified 2017-05

CONDITIONS: Development; Unilateral
Keywords: Tennis; Asymmetry; Morphological

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Humans generally develop a preferred upper and lower extremity. Due to repetitive uneven loading, this gradually results in morphological adaptations to the dominant side of the body. The corresponding morphological asymmetry can be further accentuated by (intensively) practicing a unilateral sport such as tennis, which is very popular. Yet, research on this particular topic is scarce, especially in (elite) female players. Furthermore, existing studies only examine the degree of morphological asymmetry of the upper extremity. Therefore, the aim of this study is to explore the morphological differences between the dominant and the non-dominant extremity/side on a whole body level (trunk, upper and lower extremity) in elite female tennis players.

ELIGIBILITY:
Inclusion Criteria:

* Participants will have to be professional, or elite, female tennis players.
* The players will have to participate in international tournaments in Belgium.

Exclusion Criteria:

* N/A

Ages: 16 Years to 40 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Child, Adult
Gender Based: Yes
Study Population: Professional, or elite, female tennis players
Sampling Method: Non-Probability Sample
Enrollment: 30 (Estimated)
Dates: Start 2017-07-01 (Estimated); Primary Completion 2018-12-31 (Estimated); Study Completion 2019-12-31 (Estimated)

PRIMARY OUTCOMES:
Demographics | 01/07/2017 - 31/12/2018
  Date of birth (in day/month/year to subsequently determine age) Gender: male or female Dominant upper extremity: right or left Dominant lower extremity: right or left Playing experience (in years) Average training hours (in hours per week)
  These values will be determined cross-sectionally and reported as mean and standard deviation.
Anthropometry | 01/07/2017 - 31/12/2018
  Stature (cm) Weight (kg) Body Mass Index (kg/m²) Upper extremity length (cm) Lower extremity length (cm)
  These values will be determined cross-sectionally and reported as mean and standard deviation.
Body Composition | 01/07/2017 - 31/12/2018
  1. Whole body composition: dual energy x-ray absorptiometry. Fat mass (g) lean mass (g) Bone mass (g) Bone mineral content (g) Bone mineral density (g/cm²) Bone area (cm²)
  2. Muscle thickness and subcutaneous fat layer: Ultrasound. Thickness of the subcutaneous fat (in mm) and muscle thickness (in mm) of the dominant and non-dominant M. Biceps Brachialis, M. Triceps Brachialis, M. Rectus Abdominis, M. Quadriceps Femoris and Hamstrings.
  3. Circumferences: anthropometric tape measure. Upper and lower arm (in cm) Upper and lower leg (in cm)
  These values will be determined cross-sectionally and reported as mean and standard deviation.
  In addition, all these outcome measures will be determined and reported for both the dominant and non-dominant upper and lower extremity separately.
Morphological asymmetry | 01/07/2017 - 31/12/2018
  Side-to-side difference (i.e. dominant versus non-dominant upper and lower extremity) will be calculated and expressed as a percentage (extremity symmetry index (%)) for the outcome measures described above (i.e. fat mass, muscle mass, bone mass, bone mineral content and bone mineral density).
  Extremity symmetry index = (measure dominant extremity or side / measure non-dominant extremity of side - 1) x 100

CONTACTS AND LOCATIONS:
Overall Officials: Eva D'Hondt, PhD, Study Director — Vrije Universiteit Brussel; Peter Clarys, PhD, Study Director — Vrije Universiteit Brussel
Locations (1):
- Vrije Universiteit Brussel, Brussels, Belgium

IPD SHARING:
Plan to Share IPD: No
Individual Participant Data (IPD) will not be shared or will not be available to other researchers